CLINICAL TRIAL: NCT07396480
Title: Fludarabine Plus Melphalan Versus Addition of Venetoclax to Fludarabine/Melphalan Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation in AML/MDS Patients Aged > 50 Years: a Multicenter, Randomized, Phase 3 Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJU-HSCT-VFM
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Venentoclax; Myeloid Malignancies; Conditioning; ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION; Acute Myeloid Leucemia; Myeldysplastic Syndrome (MDS)
MeSH Terms: interventions — venetoclax; fludarabine; Melphalan

STUDY DESIGN:
Intervention Model Description: 1. the Experimental Group ① Venetoclax: 400 mg/day, days -8 to -2. (Note: If fluconazole is co - administered for antifungal prophylaxis during the transplantation conditioning period, the dose of Venetoclax should be reduced to 50% of the standard dose (i.e., 200 mg/day). If voriconazole or posaconazole is used for antifungal prophylaxis, the dose of Venetoclax should be reduced to 25% of the standard dose (i.e., 100 mg/day).)
     ② Fludarabine (Flu): 30 mg/m²/day, days -7 to -3.
     ③ Melphalan (Mel) dose, adjusted according to the patient's age:
     1. For patients aged < 60 years: 140 mg/m²/day, day -2.
     2. For patients aged 60 ≤ age < 70 years: 120 mg/m²/day, day -2.
     3. For patients aged ≥ 70 years: 100 mg/m²/day, day -2.
  2. the Control Group ① Fludarabine (Flu): 30 mg/m²/day, days -7 to -3. ② Melphalan (Mel) dose, adjusted according to the patient's age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FM (Active Comparator): Fludarabine and Melphalan
  Interventions: Drug: Fludarabine and Melphalan
- VFM (Experimental): Venetoclax in combination with fludarabine and melphalan
  Interventions: Drug: Venetoclax in combination with fludarabine and melphalan

INTERVENTIONS:
Drug: Venetoclax in combination with fludarabine and melphalan — VFM Conditioning Regimen:
  1. Venetoclax: 400 mg/day, days -8 to -2. (Note: If fluconazole is co - administered for antifungal prophylaxis during the transplantation conditioning period, the dose of Venetoclax should be reduced to 50% of the standard dose (i.e., 200 mg/day). If voriconazole or posaconazole is used for antifungal prophylaxis, the dose of Venetoclax should be reduced to 25% of the standard dose (i.e., 100 mg/day).
  2. Fludarabine (Flu): 30 mg/m²/day, days -7 to -3.
  3. Melphalan (Mel) dose, adjusted according to the patient's age:
     1. For patients aged < 60 years: 140 mg/m²/day, day -2.
     2. For patients aged 60 ≤ age < 70 years: 120 mg/m²/day, day -2.
     3. For patients aged ≥ 70 years: 100 mg/m²/day, day -2.
  Arms: VFM
Drug: Fludarabine and Melphalan — FM conditioning regimen:
  1. Fludarabine (Flu): 30 mg/m²/day, days -7 to -3.
  2. Melphalan (Mel) dose, adjusted according to the patient's age:
     1. For patients aged < 60 years: 140 mg/m²/day, day -2.
     2. For patients aged 60 ≤ age < 70 years: 120 mg/m²/day, day -2.
     3. For patients aged ≥ 70 years: 100 mg/m²/day, day -2.
  Arms: FM

SUMMARY:
Allogeneic Hematopoietic Cell Transplantation (Allo-HCT) serves as a curative treatment modality for the vast majority of patients with hematological malignancies. Historically, due to the relatively high treatment-related mortality rate associated with Allo-HCT, this therapy was primarily administered to younger patients. However, the median age at onset of most hematological malignancies falls within the elderly population. For instance, the median ages at onset of Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) are 68 and 77 years, respectively. In recent years, with the advancement of transplantation techniques and the application of Reduced-intensity Conditioning (RIC) regimens, a growing number of elderly patients have undergone Allo-HCT. Data from the Center for International Blood and Marrow Transplant Research (CIBMTR) indicate that in 2017, 31% of patients who received Allo-HCT were aged over 60 years, and 6% were over 70 years old. Over the past decade, the number of elderly patients undergoing Allo-HCT has increased significantly.

Given that most elderly patients cannot tolerate conventional myeloablative conditioning regimens, RIC regimens based on Fludarabine (Flu) combined with Busulfan (Bu), or Fludarabine (Flu) combined with Melphalan (Mel) are currently widely used in elderly patients undergoing Allo-HCT. Nevertheless, the post-transplant relapse rate remains as high as 30%-55%, and the long-term GVHD-free and Relapse-free Survival (GRFS) rate fluctuates between 21% and 59%, suggesting that the efficacy of transplantation needs to be further improved. Further comparison of the commonly used RIC regimens in elderly patients-namely Flu+Bu (2-day), Flu+Bu (4-day) and Flu+Mel-has demonstrated that the Flu+Mel regimen yields superior transplantation outcomes over the Flu+Bu regimens.

At present, the optimal RIC regimen for elderly patients with hematological malignancies has not yet been clearly defined. The selection of transplantation conditioning regimens for elderly patients should strike a balance between reducing non-relapse mortality and decreasing post-transplant relapse. Over the past 20 years, an increasing number of targeted drugs acting on specific cellular signaling pathways, anti-apoptotic proteins, epigenetic regulators, and monoclonal antibodies have been introduced into clinical practice, thereby revolutionizing the treatment landscape of hematological malignancies. These novel targeted therapies not only bring hope of achieving remission to patients with hematological tumors resistant to traditional chemotherapy, but also the combined application of novel drugs and Allo-HCT is bound to fundamentally transform the overall technical system of hematopoietic stem cell transplantation. Venetoclax is a potent and selective oral inhibitor targeting the BH3 domain of the anti-apoptotic protein Bcl-2. In 2018, the FDA approved Venetoclax as a first-line induction chemotherapy agent for elderly AML patient's ineligible for intensive chemotherapy, with a complete remission rate of up to 67% and favorable tolerability¹¹. Preclinical studies using Allo-HCT animal models have confirmed that the addition of a Bcl-2 inhibitor to RIC regimens can promote donor cell engraftment, reduce the incidence of GVHD, without impairing the graft-versus-leukemia (GVL) effect¹². In recent years, clinical trials have reported the efficacy and safety of the conditioning regimen combining Venetoclax with Flu+Bu in patients with myeloid malignancies undergoing Allo-HCT. Our research center has demonstrated the favorable safety profile and promising long-term survival outcomes of the Venetoclax plus Flu+Mel conditioning regimen in a phase II clinical trial involving patients aged over 50 years with AML/MDS undergoing Allo-HCT (2024 EBMT Poster B093; 2025 EBMT Poster B126). However, the long-term superiority of this novel regimen over the conventional Flu+Mel conditioning regimen remains to be clarified.

Therefore, based on the existing findings from clinical studies and Allo-HCT animal model research, we hypothesize that incorporating Venetoclax into the Fludarabine+Melphalan conditioning regimen for elderly patients undergoing Allo-HCT is expected to improve long-term post-transplant survival and further enhance the transplantation efficacy in this patient population.

DETAILED DESCRIPTION:
Patients aged over 50 years diagnosed with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) who met the inclusion and exclusion criteria were enrolled in this study. Stratified by age (< 60 years vs. ≥ 60 years) and disease type (AML vs. MDS), the patients were randomly assigned to two groups: the control group, which received the conditioning regimen of fludarabine plus melphalan; and the experimental group, which received the conditioning regimen of venetoclax combined with fludarabine and melphalan.

1. Conditioning Regimen for the Experimental Group 1) Venetoclax: 400 mg/day, days -8 to -2. (Note: If fluconazole is co - administered for antifungal prophylaxis during the transplantation conditioning period, the dose of Venetoclax should be reduced to 50% of the standard dose (i.e., 200 mg/day). If voriconazole or posaconazole is used for antifungal prophylaxis, the dose of Venetoclax should be reduced to 25% of the standard dose (i.e., 100 mg/day).) 2) Fludarabine (Flu): 30 mg/m²/day, days -7 to -3. 3) Melphalan (Mel) dose, adjusted according to the patient's age:

   1. For patients aged < 60 years: 140 mg/m²/day, day -2.
   2. For patients aged 60 ≤ age < 70 years: 120 mg/m²/day, day -2.
   3. For patients aged ≥ 70 years: 100 mg/m²/day, day -2.
2. Conditioning Regimen for the Control Group 1) Fludarabine (Flu): 30 mg/m²/day, days -7 to -3. 2) Melphalan (Mel) dose, adjusted according to the patient's age:

   1. For patients aged < 60 years: 140 mg/m²/day, day -2.
   2. For patients aged 60 ≤ age < 70 years: 120 mg/m²/day, day -2.
   3. For patients aged ≥ 70 years: 100 mg/m²/day, day -2.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 50 years;
2. Confirmed as acute myeloid leukemia (AML) in remission prior to transplantation, high-risk myelodysplastic syndrome (MDS), or myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) by morphology, immunology, cytogenetics and molecular biology (MICM) typing;
3. Having an eligible donor and scheduled to undergo allogeneic hematopoietic stem cell transplantation (Allo-HCT) from a related or unrelated donor;
4. Karnofsky Performance Score ≥ 70;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status < 3;
6. Expected survival time > 12 weeks;
7. Voluntarily signing the informed consent form and being able to understand and comply with all study requirements.

Exclusion Criteria:

1. Complicated with severe cardiac insufficiency with a left ventricular ejection fraction (EF) < 60%; or complicated with severe arrhythmia, and assessed by the investigator as unable to tolerate the intensive conditioning regimen;
2. Complicated with severe pulmonary insufficiency (obstructive and/or restrictive ventilatory disorder), and assessed by the investigator as unable to tolerate the intensive conditioning regimen;
3. Complicated with severe liver function impairment, with liver function indicators (alanine aminotransferase [ALT], total bilirubin [TBIL]) exceeding 3 times the upper limit of normal (ULN); and assessed by the investigator as unable to tolerate the intensive conditioning regimen;
4. Complicated with severe renal insufficiency, with serum creatinine (Cr) exceeding 2 times the upper limit of normal (ULN); or with a 24-hour creatinine clearance rate (Ccr) < 50 ml/min, and assessed by the investigator as unable to tolerate the intensive conditioning regimen;
5. Suffering from severe active infection prior to transplantation, and assessed by the investigator as unable to tolerate the intensive conditioning regimen;
6. Having a history of allergic reactions or severe adverse reactions to the drugs involved in the conditioning regimen, and assessed by the investigator as ineligible for enrollment;
7. Other reasons for ineligibility assessed by the investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01-18 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
GVHD-free and Relapse-free Survival (GRFS) | 2-year
  the time from the date of transplantation to the first occurrence of any of the following events: development of grade Ⅲ-Ⅳ acute graft-versus-host disease (aGVHD); development of moderate to severe chronic graft-versus-host disease (cGVHD); disease relapse or progression; death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2-Year
  The time from the date of transplantation to death from any cause.
Progression-free Survival (PFS) | 2-Year
  The time from the date of transplantation to disease relapse, progression, or death from any cause.
Non-relapse Mortality (NRM) | 2-year
  The time from the date of transplantation to death from non-relapse causes, with disease relapse considered as a competing event.
Cumulative Incidence of Relapse (CIR) | 2-year
  Bone marrow blasts/immature cells > 5%, presence of blasts in peripheral blood, or occurrence of extramedullary leukemia; death without relapse is considered as a competing event.
Chronic Graft-versus-host Disease (cGVHD) | 2-year
  Based on the 2014 NIH Diagnostic and Grading Criteria for Chronic GVHD.
Acute Graft-versus-host Disease (aGVHD) | 100-day
  Based on the 2016 Diagnostic and Grading Criteria for Acute GVHD by Harris et al.
Immune Reconstitution (IR) | 2-year
  Recovery status of peripheral blood T, B, NK cell subsets and immunoglobulin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China